CLINICAL TRIAL: NCT05500768
Title: Efficacy of the hYpothermic Compression Bandage in the Surgical Wound of Cardiac Devices: A RAndomized Controlled Trial
Brief Title: Efficacy of the hYpothermic Compression Bandage in the Surgical Wound of Cardiac Devices
Acronym: EYRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, Head of Arrythmia Unit, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EYRA trial
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Pocket Hematoma
Keywords: cardiac devices; surgical wound; oral anticoagulation therapy; oral antiplatelet therapy; compression bandage; hypothermic therapy
MeSH Terms: conditions — Surgical Wound | interventions — Hexachlorobenzene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypothermic compression bandage (Experimental)
  Interventions: Procedure: hypothermic compression bandage
- Conventional compression bandage (Active Comparator)
  Interventions: Procedure: Conventional compression bandage

INTERVENTIONS:
Procedure: hypothermic compression bandage — a compressive bandage is applied for 8 hours to the surgical wound of the cardiac device implants, a frozen prosthesis is added
  Other Names: HCB
  Arms: hypothermic compression bandage
Procedure: Conventional compression bandage — a compressive bandage is applied for 8 hours to the surgical wound of the cardiac device implants
  Other Names: CCB
  Arms: Conventional compression bandage

SUMMARY:
The aim of this study is to evaluate the efficacy of hypothermic compression bandaging versus conventional compression bandaging, for the prevention of surgical wound hematoma of cardiac implementable electronic devices in patients undergoing chronic oral anticoagulant therapy and/or oral antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients under oral anticoagulation and/or antiplatelet treatment who were going to undergo implantation of an implanted device cardiac stimulation or generator replacement due to battery depletion

Exclusion Criteria:

* insertion of drainage in the wound,
* non-compliance with the pre-surgical antithrombotic protocol
* INR in a high therapeutic range (>3.5)
* Do not follow-up in the same hospital
* Coagulation and hemostasis disorders
* Replacement of devices due to alterations in the operation unrelated to the battery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Appearance of hematoma | 10 days
  Classification of pocket hematoma according to DeSensi et al.:
  Grade I: ecchymosis, defined as minor bleeding in the cardiac device pocket, no swelling or pain (watch and wait).
  Grade II: medium hematoma described as a palpable, bulging mass of <2cm over the implanted generator. Moderate bleeding in the pocket of the MCP or ICD, causing functional impairment or pain in the area of the heart device Grade III: severe hematoma Determined as a palpable, bulging mass >2cm. Evacuation is required if it causes tension in the skin with poor tissue perfusion, which is increasing and generates severe pain. Prolongs the patient's hospitalization or readmission for more than 24 hours. Requires immediate discontinuation of OACs or oral antiplatelets

SECONDARY OUTCOMES:
Appearance of severe hematoma | 10 days
  severe hematoma Determined as a palpable, bulging mass >2cm. Evacuation is required if it causes tension in the skin with poor tissue perfusion, which is increasing and generates severe pain. Prolongs the patient's hospitalization or readmission for more than 24 hours. Requires immediate discontinuation of OACs or oral antiplatelets

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic, Barcelona, Spain

REFERENCES:
- [Derived] Cano Valls A, Niebla M, Diago C, Domingo R, Tolosana JM, Perez S. Efficacy of Hypothermic Compression Bandages in Cardiac Device Surgical Wounds: A Randomized Controlled Trial. Adv Skin Wound Care. 2024 Sep 1;37(9):1-7. doi: 10.1097/ASW.0000000000000201. PMID 39162385